CLINICAL TRIAL: NCT03757806
Title: LiFE4D: a Home-based Physical Activity Program for Community-dwelling People With Dementia
Brief Title: Lifestyle Integrated Functional Exercise for People With Dementia: a Home-based Physical Activity Program
Acronym: LiFE4D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Collaborators: School of Health, Polytechnic Institute of Setúbal (ESS/IPS) (Unknown)
Responsible Party: Principal Investigator, Alda Sofia Pires de Dias Marques, Senior lecturer, Dr., Aveiro University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFRH/BD/120695/2016
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Dementia
Keywords: Dementia; Physical activity; Home-based; Lifestyle
MeSH Terms: conditions — Dementia; Motor Activity

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial will be conducted. Participants will be randomized to the control group or intervention group.
  The control group will receive usual care only (e.g., pharmacologic treatment), whilst the experimental group will receive an individualized home-based physical activity program at home (LiFE4D) in addition to usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive the LiFE4D in addition to usual care (e.g., pharmacologic treatment).
  Interventions: Other: Experimental group
- Control group (No Intervention): The control group will receive usual care only.

INTERVENTIONS:
Other: Experimental group — LiFE4D is an individualised programme, adapted to the participant's needs/preferences.
  People with Dementia will receive assistance to increase their physical activity multiple times/day in their everyday tasks with the support/supervision of their caregivers.
  The programme last for 12 weeks, with a lower face tracking over time with the health professional but replaced by caregivers. The intervention includes face-to-face sessions and phone calls. Face-to-face sessions aim to adapt physical activity to everyday tasks, increase tasks frequency and intensity, monitor progress, clarify doubts, motivate and manage expectations. Phone calls aim to monitor motivation/evolution and clarify doubts.
  Arms: Experimental group

SUMMARY:
Physical activity improves cognitive function and the ability to perform activities of daily living in people with dementia and reduces caregivers' burden thus, enhancing quality of life of people with dementia and their caregivers. The wish of most people with dementia, and their caregivers, is to live at their home, for as long as possible. However community-dwelling people with dementia have low levels of physical activity, increasing dependency, which often leads to institutionalization. The Lifestyle Integrated Functional Exercise (LiFE) program has been shown to decrease sedentary activity time and dependency in activities of daily living of older people, however, it has never been implemented in people with dementia. LiFE might be promising as it focuses on establishing new behaviors within selected contexts to stimulate physical activity at home. Therefore, a home-based physical activity program, based on LiFE and involving caregivers, LiFE4D, will be implemented and evaluated in community-dwelling people with dementia.

DETAILED DESCRIPTION:
Sustaining levels of regular physical activity of people with dementia is essential to maintain independence on activities of daily living, increase health-related quality of life and delay the need for institutionalization. Home-based physical activity programs, involving the caregivers, may overcome the drawbacks of the low adherence and high dropout rates by including physical activity in daily routines of people with dementia, thus increasing their motivation and confidence levels. LiFE is a home-based physical activity program which embeds training into patients' daily routines. It has shown to be well accepted and effective in healthy older people, however its effectiveness in people with dementia remains unknown.

Therefore, the primary aim of this study is to assess the impact of a home-based physical activity program, based on the LiFE program and involving the caregivers (LiFE4D), on exercise tolerance of community-dwelling people with dementia, using a randomized controlled design. The secondary aims are to:

* establish the feasibility of LiFE4D and adherence to the intervention;
* explore the impact of the LiFE4D on other health-related physical fitness components, (i.e., neuromotor, muscular strength, flexibility and body composition); physical activity, health-related quality of life, social networks and informal care time provision;
* assess the cost-effectiveness of the LiFE4D on the number of falls, healthcare resources utilization, length of hospital stay and number of respiratory infections.

To accomplish these aims, a pilot (task 1) and a randomized controlled study (task 2) will be conducted. LiFE4D will be centered on the duo participant/caregiver capacities and potentialities and it will be a significant contribution towards the development and implementation of an innovative home-based physical activity intervention. Additionally, it will inform the cost-effectiveness of this intervention in people with dementia. Ultimately, findings from this project will provide guidance to national and international health policies on physical activity promotion in community-dwelling people with dementia.

Task 1: LiFE4D - Pilot study

A pilot study will inform sample size, recruitment/randomization procedures and feasibility of LiFE4D.

Ethical approval will be obtained from Ethics and Data Protection Committees. People with dementia will be included if they: have a diagnosis of mild/moderate dementia according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V); are living at home; are not participating in exercise training; are able to follow instructions and have a caregiver. People with dementia will be excluded if they: have been hospitalized in the previous month; present any clinical condition that precludes them to be involved in physical activity; have been taking medication that affect exercise capacity/bone density. Eligible participants will be identified via care homes, day care centers and Alzheimer Cafes (meetings with people with dementia and families). These institutions will contact eligible participants. Informed consent will be obtained from interested people with dementia and legal representatives.

The Experimental Group (EG) will receive the LiFE4D in addition to usual care (e.g., pharmacologic treatment), whilst the Control Group (CG) will receive usual care only.

Protocol will take approximately 1h and data will be collected at participants' home at baseline and after 12 weeks. ActiGraph will be used during one week before and one week after the 12 weeks. Participants will wear the ActiGraph for at least 6 consecutive days. Additionally, at baseline the EG group will be assessed (with observation and a structured questionnaire) on their daily routines to adjust the intervention to each participant's needs.

Feasibility measures. Adherence to LiFE4D and number/reasons of dropouts will be collected.

Intervention LiFE4D information will be offered during a collective session for the EG, i.e., people with dementia and their caregivers. Then, the individualized program will be set up, adapted to the participant's needs/preferences.

People with dementia will train balance, flexibility, endurance and strength multiple times/day in their everyday tasks with the support/supervision of their caregivers. Strategies to improve balance include "reduce base of support" (e.g., working at the kitchen while standing on one leg), "move to limits of sway", "shift weight from foot to foot", "step over objects" and "turning and changing direction". Strategies to increase strength and endurance include "bend your knees" (e.g., squatting instead of bending at the waist to close a drawer or to picking things up from the floor), "on your toes", "up the stairs", "on your heels", "sit to stand", "walk sideways" and "tighten muscles". Intensity of training will be adjusted throughout the program based on the regular evaluation of balance and strength.

The program will last for 12 weeks, with a lower face tracking over time with the health professional but replaced by involvement of caregivers. Specifically includes:

* Weeks 1-4: 3 face-to-face sessions/week;
* Weeks 5-8: 2 face-to-face sessions/week and a biweekly phone call;
* Weeks 9-11: 1 face-to-face session/week and a phone call;
* Week 12: 1 phone call. Face-to-face sessions aim to adapt physical activity to everyday tasks, increase tasks frequency and/or intensity, monitor progress, clarify doubts, motivate higher daily energy expenditure and manage expectations. Telephone contacts aim to monitor people with dementia's motivation/evolution and clarify doubts of people with dementia and caregivers.

Task 2: Implementation and evaluation of LiFE4D

Informed by task 1, a powered (80%, alpha=0.05) randomized controlled trial will be designed.

Data collection times: as described in task 1, however, additional assessments for follow up will be conducted at 3, 6 months after the LiFE4D, to assess short- and long-term results.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of mild/moderate dementia according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V); are living at home; are not participating in exercise training; are able to follow instructions and have a caregiver.

Exclusion Criteria:

* have been hospitalized in the previous month; present any clinical condition that precludes them to be involved in physical activity; have been taking medication that affect exercise capacity/bone density.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
2 Minute Step test - change in exercise tolerance | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  Participants' exercise tolerance will be assessed with the 2 Minute Step Test, counting the number of times the right knee is raised to the level of the mark on the wall or board (half way between the participant's knee and iliac crest). Higher number of repetitions indicate better performance.

SECONDARY OUTCOMES:
Addenbrooke's Cognitive Examination III - change in cognitive function | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  The Addenbrooke's Cognitive Examination III is a brief cognitive measure that assesses five cognitive domains: attention, memory, verbal fluency, language and visuospatial abilities. This measure's score ranges between 0-100 points with higher scores indicating better cognitive function.
Brief Balance Evaluation System Test - change in balance | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  The Brief Balance Evaluation System Test (Brief-BESTest) is a 6 item measure that assesses 6 balance domains: biomechanical constraints, stability limits/verticality, anticipatory postural responses, postural responses, sensory orientation, and stability in gait. The Brief-BESTest has a total score of 24 points and higher scores indicate better performance.
Brief Physical Activity Assessment tool - change in self-reported physical activity | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  Participants' self-reported physical activity will be assessed with the Brief Physical Activity assessment tool. This measure consists of 2 questions assessing the frequency and duration of intense and moderate physical activity undertaken in a usual week. A total score was calculated (range 0-8), in which higher scores correspond to higher physical activities levels.
Accelerometer-based activity monitors - change in physical activity levels | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  Physical activity levels will be collected with the activity monitors GT3X+ (ActiGraph) to measure the number of steps/day and daily energy expenditure during one week.
Handgrip Dynamometer - change in maximum isometric strength of the hand and forearm muscles | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  Participants' hand and forearm strength will be collected with the Handgrip Dynamometer that measures muscular strength in kilograms (0-90) of the maximum prehension.
30 second sit to stand test - change in lower limb strength | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  Participants' lower limb strength will be collected with the 30 second sit to stand test, that consists into sit and stand as many time as possible during 30 seconds. Higher number of repetitions indicate better performance.
Grocery Shelving Task - change in upper limb functionality | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  Participants' upper limb functionality will be collected with the Grocery Shelving Task (GST). The GST consists of place twenty 420-g grocery cans (placed in 2 shopping bags) on a shelf (15 cm above shoulder level in the standing position), with a 90 cm table placed 30 cm in front of the shelf, as quickly as possible. Lower time to perform the task indicate better performance.
Chair sit and reach test - change in flexibility | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  The Chair Sit and Reach test measures the distance between the tip of the fingers and the toes on a sat position. If the participant do not reach the toes has a negative score (cm) and, if overlap has a positive score (cm), with higher scores indicating better performance.
Functional Reach Test - change in functionality | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  Functional Reach Test assesses the distance reached forward by the participants, without taking a step, on a standing position. Higher scores indicate better performance.
Timed Up and Go test - change in functional mobility | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  The Timed Up and Go test consists in counting the time (seconds) to raise from a chair, walk 3 meters at a comfortable pace, turn, walk back and seat on the chair. Lower time indicate better performance.
Physical Performance Test - change in overall functionality | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  The Physical Performance Test assesses multiple domains of physical function using tasks that simulate activities of daily living. This measure has 9-items with a total score of 36 points, with higher scores indicating better performance.
Peak Flow Meter - change in lung function | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  Participants' lung function will be collected with the Peak Flow Meter equipment that measures the peak expiratory flow (MicroPeak, CareFusion, Basingstoke, United Kingdom - Standard range, EU (EN 23747) scale). Higher scores indicate better performance.
Maximal inspiratory (MIP) and expiratory (MEP) pressures and Sniff Nasal Inspiratory Pressure (SNIP) - change in respiratory muscle strength | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  Participants' respiratory muscle strength will be collected using a respiratory pressure gauge (MicroRPM, CareFusion, Kent, United Kingdom) that measures maximal inspiratory and expiratory pressures and sniff nasal inspiratory pressure. Higher values indicate better performance.
Quality of Life in Alzheimer's Disease scale - change in health-related quality of life | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  Participants' health-related quality of life will be collected using the Quality of Life in Alzheimer's Disease scale (QoL-AD), that is an interview format scale. The QoL-AD has 13 items with a total score of 52 points, with higher scores indicating better performance.
Short Form Zarit Burden Interview - change in caregivers' burden | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  Caregivers' burden will be collected using the Short Form Zarit Burden Interview scale, with 12 items and a total score range 0-48 points. Higher scores indicate higher burden.
Resource Utilization in Dementia - Lite - change in informal time provision | Assessment at baseline, post (3 months) and 3 months and 6 months follow-up for experimental and control groups.
  Informal time provision will be collected using the Resource Utilization in Dementia - Lite (RUD-Lite) questionnaire. This questionnaire is not scored, it provides information, such as, hospitalizations, time spent assisting with personal ADLs, time spent supervising the participant, social services.

CONTACTS AND LOCATIONS:
Overall Officials: Alda S Marques, PhD, Principal Investigator — School of Health Sciences of the University of Aveiro (ESSUA)
Locations (1):
- University of Aveiro, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No